CLINICAL TRIAL: NCT05336214
Title: PRimary Care Education and Practice Adoption Resource Evaluation for Continuous Glucose Monitoring
Brief Title: Implementing Continuous Glucose Monitoring in Primary Care for Patients With Diabetes
Acronym: PREPARE4CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-4269
Record Dates: First submitted 2022-03-23; First posted 2022-04-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Refer (Experimental): Practice referral of patients to a virtual CGM initiation service
  Interventions: Other: Virtual CGM initiation service
- Learn (Experimental): Practice completion of online educational module, American Academy of Family Physicians (AAFP) Transformation in Practice Series (TIPS) on continuous glucose monitoring in primary care
  Interventions: Other: Online educational module on CGM
- Learn + Practice Facilitation (Experimental): Practice completion of online educational module, American Academy of Family Physicians (AAFP) Transformation in Practice Series (TIPS) on continuous glucose monitoring in primary care plus practice facilitation
  Interventions: Other: Online educational module on CGM; Other: Practice facilitation

INTERVENTIONS:
Other: Virtual CGM initiation service — Primary care practices will refer patients to an external virtual initiation service staffed by clinical pharmacists, diabetes care and education specialists, and physicians. The initiation service will communicate with eligible patients (referred to the virtual initiation service by their provider) to review device options and provide patient education and support on device use for up to 12 months to help initiate use of the device. The initiation service will communicate with a patient's provider about treatment and follow up, but will not make treatment recommendations directly to patients.
  Arms: Refer
Other: Online educational module on CGM — Primary care practices will complete online educational modules, the American Academy of Family Physicians Transformation in Practice Series on CGM. This series includes education on diabetes; glucose monitoring; evidence behind CGM; CGM implementation tools, strategies, and workflows; billing, reimbursement, and insurance authorization of CGM; and tools and strategies to use CGM for quality improvement in diabetes care.
  Arms: Learn; Learn + Practice Facilitation
Other: Practice facilitation — A practice facilitator will support primary care practices in training team members using the American Academy of Family Physicians Transformation in Practice Series on CGM and in implementation of strategies to support CGM use for patients with diabetes in primary care.
  Arms: Learn + Practice Facilitation

SUMMARY:
The overarching goal of this study is to decrease disparities and increase access to continuous glucose monitoring (CGM) for patients with diabetes, regardless of where people receive their diabetes care. This study aims to evaluate the effectiveness of three implementation strategies for CGM in primary care practices in an efficient, sustainable, and scalable fashion. The investigators will also perform economic analysis of the implementation strategies.

This 3-year study will compare practices that implement CGM with (a) an evidence-based educational module only, (b) an educational module plus practice facilitation support, or (c) a virtual CGM initiation clinic for patients. There will be up to 30 practices in each group for a possible total of 90 primary care practices. The investigators expect to enroll up to 500 patient participants across these 90 practices and to compare outcomes among patients from each study arm.

This comparison will help investigators to understand the different implementation strategies and their ability to help primary care practice adopt, implement, and maintain CGM for their patients. The information the investigators collect will also help to understand how patients in these primary care practices experience initiation and use of CGM. The results will help to develop strategies and tools to train more primary care practices to offer CGM more widely to patients for whom it is recommended, especially for those where access to specialty care is limited.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 and 89 years
* Has diagnosis of type 1 diabetes or type 2 diabetes
* Recommended by primary care clinician to use continuous glucose monitoring to manage diabetes
* Ability to read or speak English or Spanish

Exclusion Criteria:

* Pregnant women
* Younger than 18 years of age
* Older than 89 years of age

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in practice-reported prescriptions of Continuous Glucose Monitors | Baseline, 6, and 12 months from baseline
  Change in number of patients over time by study arm with diabetes prescribed a Continuous Glucose Monitoring Device. This is a practice-level indicator of patient reach in primary care settings.

SECONDARY OUTCOMES:
Glycemic control (a) | Baseline to 12 months after enrollment
  Change in HbA1c over time by study arm.
Glycemic control (b) | Baseline, 3, 6, and 12 months from baseline
  Change in Time in Range for each participant based on Continuous Glucose Monitor recordings (past 10-14 days), by study arm
Glycemic control (c) | Baseline, 3, 6, and 12 months from baseline
  Change in Time above range for each participant with various glycemic ranges based on Continuous Glucose Monitor recordings (past 10-14 days), by study arm
Glycemic control (d) | Baseline, 3, 6, and 12 months from baseline
  Change in Time below range for each participant with various glycemic ranges based on Continuous Glucose Monitor recordings (past 10-14 days), by study arm
Glycemic control (e) | Baseline, 3, 6, and 12 months from baseline
  Change in GMI (glucose management indicator) for each participant based on Continuous Glucose Monitor recordings (past 10-14 days), by study arm
Diabetes-related distress | Baseline, 3, and 6 months from baseline
  Change in diabetes-related distress over time by study arm, as measured by the Diabetes Distress Screening Scale (DSS). This is a patient-level indicator measuring dimensions of emotional burden and regimen-related distress; changes in distress metrics are expected as an outcome of increased Continuous Glucose Monitor prescriptions. Ratings are averaged across the 17 scale items for a DSS score ranging between 1 and 6. Higher scores indicate greater distress (worse outcome), with a score of 3 or greater indicating "moderate distress."
Glucose Monitoring Satisfaction Survey | Baseline, 3, and 6 months from baseline
  Change in Patient device satisfaction over time by study arm, as measured by the Glucose Monitoring System Satisfaction Survey (GMSS). This is a patient-level indicator measuring dimensions of emotional burden and regimen-related distress; changes in distress metrics are expected as an outcome of increased CGM prescriptions. Ratings are averaged across scale items for a GMSS score ranging between 1 and 5. Higher scores indicate greater satisfaction (positive outcome).
Cost Analysis and Economic Sustainability | 6 months from baseline
  Counts of Current Procedural Terminology (CPT)/Healthcare Common procedure Coding System (HCPCS) codes collected for all visits with Continuous Glucose Monitor patients and calculated using the Medicare Reimbursement Rate
Implementation and Maintenance | 6 and 12 months from baseline
  The Implementation Milestones Checklist will allow the investigators to identify differences between study arms' ability to meet and/or maintain various steps in the intervention timelines. This is a practice-level indicator of ability to sustain the intervention and any positive effects. Items are averaged for an overall measure of practice implementation, with ratings ranging from 0 (Don't plan to use) to 4 (completed). Higher scores indicate greater implementation (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Oser, MD, Principal Investigator — University of Colorado Denver | Anschutz Medical Campus; Sean Oser, MD, MPH, Principal Investigator — University of Colorado Denver | Anschutz Medical Campus
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiggins KT, Hall TL, Jortberg B, Dickinson WP, Dickinson LM, Parascando JA, Fernald DH, Sobczak C, Oser SM, Oser TK. Primary care practices' choice of implementation strategy for continuous glucose monitoring for patients with diabetes: a multiple methods study within a larger hybrid type-3 effectiveness-implementation study. BMC Prim Care. 2025 Jun 9;26(1):195. doi: 10.1186/s12875-025-02903-0. PMID 40490741